CLINICAL TRIAL: NCT05258669
Title: A Phase 2/3, Observer-Blind, Immuno-bridging, and Broadening Study of a Whole, Inactivated Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV-2) Vaccine (BBV152) in Healthy Adults
Brief Title: Immuno-bridging and Broadening Study of a Whole, Inactivated COVID-19 Vaccine BBV152 in Healthy Adults
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ocugen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OCU-002
Record Dates: First submitted 2022-02-22; First posted 2022-02-28 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — BBV152 COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: 1:1 randomization ratio
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An unblinded pharmacist or another qualified individual will prepare and provide the syringe in a blinded manner to the study vaccine administrator (a trained and qualified study nurse, medical doctor, or otherwise qualified health care professional) who will perform the injection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BBV152 (Active Comparator): BBV152
  Interventions: Biological: BBV152
- Placebo (Placebo Comparator): 0.9% normal saline
  Interventions: Biological: BBV152

INTERVENTIONS:
Biological: BBV152 — Each participant will receive 2 doses of the investigational product intramuscular injection of either 6 μg of BBV15 vaccine or placebo.
  Other Names: Covaxin

SUMMARY:
A randomized, observer-blind, placebo-controlled immuno-bridging, and broadening study to demonstrate the equivalence of the immune response between participants enrolled in Phase 3 efficacy trial in India and demographically diverse healthy adult participants in the US which matched in age and vaccine formulation setting to whom those efficacy results are extrapolated; and to assess the broadening of the BBV152 in participants who previously received two shots of messenger ribonucleic acid (mRNA) COVID-19 vaccine at least 6 months earlier or one-shots of viral vector J&J/Janssen COVID-19 vaccine at least 2 months earlier. Safety and tolerability evaluation is a secondary endpoint.

DETAILED DESCRIPTION:
Participants in stable health will be randomly assigned into one of four groups based on their age to receive either 6 µg of BBV152 or placebo in a 1:1 ratio. Each participant will receive 2 doses of the study vaccine by 0.5 mL intramuscular injection, the first on Day 0 and the second on Day 28. Data will be collected in an observer-blind manner.

Safety will be monitored by the Data and Safety Monitoring Board. The Data and Safety Monitoring Board will convene to perform safety reviews at 2 and 6 months and for immediate concerns regarding safety observations as needed.

Safety assessment will include monitoring solicited, unsolicited, serious, medically attended adverse events and potentially immune medicated medical conditions.

Since this is a bridging study, the maximum sample size of the data from the previous study will be 31 samples from the <65 years population and 358 with samples from the 18 to <65 years population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥ 18 years of age at the time of informed consent.
2. The participant is capable of providing signed informed consent.
3. The participants who consent, are willing and able to comply with all scheduled visits, treatment plans, laboratory tests, lifestyle considerations, and other study procedures.
4. Have negative the Cue™ SARS-CoV-2 Test of anterior nasal specimens.
5. Participants must have received two documented doses of mRNA vaccine a minimum of 180 days from their last dose prior to enrollment or One documented dose of viral vector J&J/Janssen COVID-19 vaccine a minimum 60 days from their dose prior to enrollment, or A documented dose of the booster shot of the mRNA COVID-19 vaccine (Comirnaty or Spikevax) a minimum of 150 days from their last dose prior to enrollment, or No vaccination history of COVID-19 vaccine and no history of COVID-19 disease (self-report, on-site inquiry).
6. The participant must agree not to take the influenza vaccine until 30 days after the second dose of vaccination and not take any other vaccines for the entire duration of the study.
7. Participants must be in relatively stable health based on the site Investigator's judgment, as determined by medical history, physical examination, and the following criteria:

   1. Stable health for age (defined as no new conditions per medical history, new medications in a different therapeutic class, or change in a daily dose of existing prescription medications within the 45 days preceding Screening).
   2. Participants may be on chronic or as-needed medications if, in the opinion of the Investigator, these pose no additional risk to participant safety or assessment of reactogenicity, and immunogenicity and their use is not for management of a worsening of medical diagnosis or condition.
8. Participants are expected to be available for the duration of the study and can be contacted by telephone during study participation.
9. Have a non-clinically significant 12-lead ECG
10. Participants must be healthy based on clinical laboratory tests performed at screening.
11. Female participants of childbearing potential may be enrolled in the study if the participant fulfills all the following criteria:

    * Has a negative urine pregnancy test at Screening and prior to each study dose
    * Has agreed to continue adequate contraception through 3 months following the second dose of the IP
    * Has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first dose (Day 0)
    * Is not currently breastfeeding Adequate female contraception is defined as consistent and correct use of a Food and Drug Administration (FDA) approved contraceptive method in accordance with the product label.
12. Male participants engaging in activity that could result in the pregnancy of sexual partners must agree to practice adequate contraception and refrain from sperm donation from the time of the first dose and through 6 months after the second dose.

Adequate contraception for male participants is defined as:

* Monogamous relationship with a female partner using an intrauterine device or hormonal contraception (described above)
* Use of barrier methods and spermicide Male participants with partners who have become pregnant prior to Screening are eligible to participate in the study.

  15. Have a body mass index (BMI) less than 35.0 kg/m2 at Screening.

Exclusion Criteria:

1. History of COVID-19 disease (self-report, on-site inquiry).
2. Presence of fever or other acute illness at the time of enrollment. Fever is defined as an oral temperature ≥ 38.0°C/100.4°F.
3. History or current clinically significant cardiac disease, such as myocarditis, pericarditis, ventricular arrhythmia requiring therapy, uncontrolled hypertension, or any history of symptomatic congestive heart failure (CHF).
4. Has significant renal, vascular, pulmonary, gastrointestinal, neurologic, hematologic, rheumatologic, oncologic, psychiatric disease, or immune-deficiency or other medical disorders not excluded by other exclusion criteria, which, in the opinion of the Investigator, may either put the individual at risk because of participation in the study or influence the safety or the volunteer's ability to participate in the study.
5. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g., anaphylaxis) to any component of the study intervention(s).
6. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
7. History of autoimmune disease or an active autoimmune disease requiring therapeutic intervention, including but not limited to systemic lupus erythematosus (e.g., rheumatoid arthritis, polyarticular juvenile idiopathic arthritis, psoriatic arthritis, ankylosing spondylitis, multiple sclerosis, systemic lupus erythematosus)
8. Has bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the Investigator, contraindicate intramuscular injection.
9. Receipt of treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids (equivalent to prednisone ≥ 10mg/day for the duration of ≥ two weeks), e.g., for cancer or an autoimmune disease, or planned receipt throughout the study period. If systemic corticosteroids have been administered short-term (<14 days) for treatment of an acute illness, participants should not be enrolled in the study until corticosteroid therapy has been discontinued for at least 28 days (about 4 weeks) before study intervention administration.
10. Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, from 60 days (about 2 months) before study intervention administration, or receipt of any passive antibody therapy specific to COVID-19 from 90 days (about 3 months) before study intervention administration or planned receipt throughout the study.
11. Has participated in an interventional clinical trial within the 4 weeks prior to randomization.
12. Known sensitivity to any components of the study vaccine.
13. The participant has received the influenza vaccine within 14 days prior to enrollment and any other vaccine within 28 days prior to randomization.
14. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IP.
15. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody. Participants who have been effectively treated for hepatitis C, as evidenced by a negative hepatitis C ribonucleic acid (RNA) confirmation test and who no longer require antiviral therapy, are eligible for participation.
16. Known or suspected history of alcohol or Drug Enforcement Administration (DEA) Schedule 1 (including for cannabis, even where legal) or excessive intake of alcohol as judged by the Investigator. Benzodiazepines for anxiety disorders and stimulants for attention deficit hyperactivity disorder are not exclusionary if the participant has been on a stable dose for more than 3 months prior to Screening and each study dosing and if the participant can produce a valid, current prescription for the medication. Propoxyphene, opioids, or combinations containing these medications (including as used for opioid addiction) are not permitted regardless of prescription status. Note: A positive Screening urine drug screen may not be repeated.
17. Donated blood products within the 4 weeks prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Compare immune response measured by serum neutralizing antibodies against Wild-Type SARS-CoV-2 in US-based participants and age-matched controls participants who participated in the Phase 3 efficacy trial in India. | Vaccination days (Day 0 and Day 28), Day 56 and Day 84
  Serum neutralizing antibodies against Wild-Type SARS-CoV-2 will be measured by Microneutralization Test (MNT) assay.

SECONDARY OUTCOMES:
Evaluate the change over time in immunogenicity of two doses of BBV152 measured by MNT neutralizing antibodies. | Day0, Day 28, Day 56 and Day 84
  * Geometric Mean Titer (GMT) as measured by MNT neutralizing antibodies against Wild-Type and Omicron and ELISA Immunoglobulin G (IgG) Abs against Spike, Receptor-Binding Domain (RBD), and N protein in BBV152 treatment group, overall, and stratified by age group.
  * Geometric Mean Fold Rises (GMFR) as measured by MNT neutralizing antibodies against Wild-Type and Omicron and ELISA IgG Abs against Spike, RBD, and N protein in BBV152 treatment group, overall, and stratified by age group.
  * Geometric Mean Titer, Geometric Mean Fold Rises, and Seroconversion rate as measured by MNT nAbs against Omicron at Day 0, Wild Type at Day 0 and Day 56 and ELISA IgG Abs against Spike, RBD, and N protein at Day 0, Day 28, Day 56, Day 84 in the placebo treatment group.
Evaluate the immunogenicity of two doses of BBV152 measured by MNT neutralizing antibodies. | Day 0, Day 28, Day 56 and Day 84
  * Geometric Mean Titer (GMT) as measured by MNT Neutralizing Antibodies (nAbs) against Wild-Type and Omicron and ELISA IgG Abs against Spike, RBD, and N protein in BBV152 treatment group, overall, and stratified by age group.
  * Geometric Mean Fold Rises (GMFR) as measured by MNT nAbs against Wild-Type and Omicron and ELISA IgG Abs against Spike, RBD, and N protein in each BBV152 treatment group, overall, and stratified by age group.
  * Geometric Mean Titer, Geometric Mean Fold Rises, and Seroconversion rate as measured by MNT nAbs against Omicron at Day 0, Wild Type at Day 0 and Day 56 and ELISA IgG Abs against Spike, RBD, and N protein at Day 0, Day 28, Day 56, Day 84 in the placebo treatment group.
Evaluate the serious adverse events (SAEs) | 1 year
  Total count, duration, frequency of participants, and proportion of participants reporting serious adverse events (SAEs)
Evaluate response rate of anti-SARS-CoV-2 IgG antibody seroconversion from negative to positive following 28 days of BBV152 administration | Day 0, Day 28, Day 56 and Day 84
  * Seroconversion rate, defined as 4-fold rise from day 0, at days 28, 56, and 84 as measured by MNT neutralizing antibodies against Wild-Type and Omicron and ELISA IgG Abs against Spike, RBD, and N protein in BBV152 treatment group, overall, and stratified by age group.
  * Seroconversion rate as measured by MNT nAbs against Omicron at Day 0, Wild Type at Day 0 and Day 56 and ELISA IgG Abs against Spike, RBD, and N protein at Day 0, Day 28, Day 56, Day 84 in the placebo treatment group.
Evaluate the immunogenicity of the single dose of BBV152. | Day 0, Day 28, Day 56 and Day 84
  * Geometric Mean Titer (GMT) as measured by MNT neutralizing antibodies against Wild-Type and Omicron and ELISA IgG Abs against Spike, RBD, and N protein in BBV152 treatment group, overall, and stratified by age group.
  * Geometric Mean Fold Rises (GMFR) as measured by MNT neutralizing antibodies against Wild-Type and Omicron and ELISA IgG Abs against Spike, RBD, and N protein in BBV152 treatment group, overall, and stratified by age group.
  * Geometric Mean Titer, Geometric Mean Fold Rises, and Seroconversion rate as measured by MNT nAbs against Omicron at Day 0, Wild Type at Day 0 and Day 56 and ELISA IgG Abs against Spike, RBD, and N protein at Day 0, Day 28, Day 56, Day 84 in the placebo treatment group.
Evaluate immune-broadening, as measured by MNT neutralizing antibodies, compare the sera taken from previously mRNA or viral vector vaccinated US-based participants with sera taken from previously mRNA or Viral Vector vaccinated placebo controls. | Day 0, Day 28, Day 56 and Day 84
  * Geometric Mean Titer (GMT) as measured by MNT neutralizing antibodies against Wild-Type and Omicron and ELISA IgG Abs against Spike, RBD, and N protein in BBV152 treatment group, overall, and stratified by age group.
  * Geometric Mean Fold Rises (GMFR) as measured by MNT neutralizing antibodies against Wild-Type and Omicron and ELISA IgG Abs against Spike, RBD, and N protein in BBV152 treatment group, overall, and stratified by age group.
  * Geometric Mean Titer, Geometric Mean Fold Rises, and Seroconversion rate as measured by MNT nAbs against Omicron at Day 0, Wild Type at Day 0 and Day 56 and ELISA IgG Abs against Spike, RBD, and N protein at Day 0, Day 28, Day 56, Day 84 in the placebo treatment group.
Evaluate the medically attended adverse events (MAAEs). | 1 year
  Total count, duration, frequency of participants, and proportion of participants reporting medically attended adverse events (MAAEs)
Evaluate potential immune-mediated medical conditions (PIMMCs). | 1 year
  Total count, duration, frequency of participants, and proportion of participants reporting potential immune-mediated medical conditions (PIMMCs)
Evaluate the adverse events of special interest (AESI). | 1 year
  Total count, duration, frequency of participants, and proportion of participants reporting adverse events of special interest (AESI).
Evaluate the unsolicited adverse events. | 28 days following the first vaccination and 1 year following the last dose of vaccination
  Total count, duration, frequency of participants, and proportion of participants reporting unsolicited adverse events.
Evaluate the solicited adverse events. | for 7 days following each dose of vaccination
  Total count, frequency of participants, and proportion of participants solicited local and systemic adverse events.

OTHER OUTCOMES:
Explore cell based immune response in a subset of participants following 28 days of the second dose of BBV152 administration | D0 and Day 56
  * Geometric Mean Titer (GMT) as measured by MNT neutralizing antibodies against Wild-Type and Omicron and ELISA Immunoglobulin G (IgG) Abs against Spike, Receptor-Binding Domain (RBD), and N protein in the BBV152 treatment group and a subset of the placebo treatment group, overall, and stratified by age group.
  * Geometric Mean Fold Rises (GMFR) as measured by MNT neutralizing antibodies against Wild-Type and Omicron and ELISA IgG Abs against Spike, RBD, and N protein in the BBV152 treatment group and a subset of the placebo treatment group, overall, and stratified by age group.
Explore the immunogenicity of one and two doses of BBV152 against future variants of concern. | Day0, D28, and Day 56
  * Geometric Mean Titer (GMT) as measured by MNT neutralizing antibodies against Wild-Type and Omicron and ELISA Immunoglobulin G (IgG) Abs against Spike, Receptor-Binding Domain (RBD), and N protein in BBV152 treatment group and a subset of the placebo treatment group, overall, and stratified by age group.
  * Geometric Mean Fold Rises (GMFR) as measured by MNT neutralizing antibodies against Wild-Type and Omicron and ELISA IgG Abs against Spike, RBD, and N protein in the BBV152 treatment group and a subset of the placebo treatment group, overall, and stratified by age group.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Qamar, MD, MPH, CMI, Study Director — Ocugen
Locations (10):
- United States (10):
  - Voyage Medical, Tempe, Arizona
  - Angels Clinical Institute, Miami, Florida
  - Suncoast Research Group LLC, Miami, Florida
  - Palm Springs Community Health Center, Miami Lakes, Florida
  - Clinical Site Partners, Winter Park, Florida
  - IACT Health, Columbus, Georgia
  - Jay Meyer Meridian Research, Lincoln, Nebraska
  - PRX Research, Dallas, Texas
  - Wellness Clinical Research, McKinney, Texas
  - Meridian Research 3235 Academy Ave, Portsmouth, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Non-Human Primate Efficacy Study Immunogenicity and protective efficacy of inactivated SARS-CoV-2 vaccine candidate, BBV152 in rhesus macaques — https://www.nature.com/articles/s41467-021-21639-w
- See also: Neutralization of Brazil variant of concern P2 (B.1.1.28) Neutralization of B.1.1.28 P2 variant with sera of natural SARS-CoV-2 infection and recipients of BBV152 vaccine — https://www.biorxiv.org/content/10.1101/2021.04.30.441559v1